CLINICAL TRIAL: NCT01460953
Title: Use of a Training Video to Teach Medical Students About Health Literacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Cliff Coleman, Assistant Professor of Family Medicine, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OHSU IRB00007828
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Health Literacy
Keywords: curriculum; training; Medical student Knowledge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- training intervention (Experimental): Students participating in didactic training
  Interventions: Behavioral: health literacy training video

INTERVENTIONS:
Behavioral: health literacy training video — participants will watch a training video

SUMMARY:
1. Briefly describe the purpose of this protocol: This study is designed to evaluate the effectiveness of an educational training video on the topic of health literacy for medical students.
2. Briefly summarize how participants are recruited: OHSU medical students attending mandatory trainings on the topic of health literacy during the 1st and 2nd years of medical school will be invited to participate in the study.
3. Briefly describe the procedures subjects will undergo: Completion of a short self-administered anonymous survey before and after viewing a 23-minute video about health literacy.
4. If applicable, briefly describe survey/interview instruments used: A 12-item pre-test questionnaire and 13-item post-test questionnaire designed to assess individuals' knowledge about health literacy, and intended clinical practices with respect to health literacy.
5. If this is a clinical trial using an experimental drug and/or device, or an approved drug and/or device used for an unapproved purpose, briefly describe the drug and/or device: n/a
6. Briefly describe how the data will be analyzed to address the purpose of the protocol: Demographics and responses to individual items will be reported as frequencies and percentages within the sample. The investigators will use a chi-square analysis to stratify responses by demographic groups and t-tests to measure possible changes over time.

ELIGIBILITY:
Inclusion Criteria:

* 1st-year medical student at OHSU

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in knowledge | immediately following the intervention, and at 12-month follow-up
  The investigators will measure knowledge about health literacy before and after an educational intervention

CONTACTS AND LOCATIONS:
Overall Officials: Clifford A Coleman, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU School of Medicine, Portland, Oregon, United States